CLINICAL TRIAL: NCT01317589
Title: Treatment of Pain in Head-and-Neck Cancer Patients: is Methadone More Effective Than Fentanyl?
Brief Title: Treatment of Pain in Head-and-Neck Cancer Patients: is Methadone More Effective?
Acronym: 310111-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 11-2-007
Record Dates: First submitted 2011-02-16; First posted 2011-03-17 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pain; Cancer of Head and Neck
Keywords: Pain; Cancer of Head and Neck; methadone; Fentanyl
MeSH Terms: conditions — Pain; Head and Neck Neoplasms | interventions — Fentanyl; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl (Active Comparator): active pain treatment with fentanyl patch
  Interventions: Drug: fentanyl
- methadone (Experimental): active pain treatment with methadone
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: fentanyl — T = 0
  * start methadone 2 x 2,5 mg or fentanyl patch 12 μg/uur
  * breakthrough medication: 50 µg fentanyl nose spray or fentanyl stick 400 µg till 6x/day
  T=1
  1 week
  * if necessary increase dose strong opioid with 50%
  T=2 3 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  T=3 5 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  T = 4 9 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  Other Names: Durogesic
  Arms: fentanyl
Drug: methadone — T = 0
  * start methadone 2 x 2,5 mg or fentanyl patch 12 μg/uur
  * breakthrough medication: 50 µg fentanyl nose spray or fentanyl stick 400 µg till 6x/day
  T=1
  1 week
  * if necessary increase dose strong opioid with 50%
  T=2 3 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  T=3 5 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  T = 4 9 weeks
  * if necessary increase dose strong opioid with 50%
  * if necessary decrease dose strong opioid with 30%
  Other Names: Symoron
  Arms: methadone

SUMMARY:
Background of the study:

Treatment of Pain in Head-and-Neck Cancer Patients:

is methadone more effective than fentanyl?

Pain is a prevalent symptom in patients with cancer. A neuropathic component is seen in one third of the patients. In patients with head-and-neck cancer neuropathic pain is far more prevalent than in a general cancer population: 46-64%. Treatment of neuropathic pain is complex and available treatment modalities achieve (partial) pain relief in only 40-60% of patients. The N-Methyl-D-Aspartate Receptor (NMDAR) plays a central role in the mediation of neuropathic pain. NMDAR blockers could be a new approach to treat neuropathic pain in patients with cancer.

Methadone is a strong opioid but at the same time significant non-competitive NMDA-receptor antagonist qualities have been described. Many small studies and case-reports describe the successful rotation from different strong opioids to methadone. There are no studies that selected patients with (predominantly) neuropathic pain to be treated with methadone, whereas this group of patients is expected to profit from the NMDAR-antagonist properties of methadone.

Objective of the study:

This randomised controlled trial (RCT) aims to investigate whether addition of a NMDAR-antagonist to a strong opioid (methadone) is superior in the treatment of predominantly neuropathic pain over a strong opioid alone (fentanyl) in terms of pain relief and time to achieve significant pain relief.

Study design:

Open label randomised controlled trial

Study population:

opioid naïve patients with histological proven head-and-neck cancer and (partly) neuropathic pain with a NRS score of ≥ 4, age =/> 18 years

Intervention Treatment with methadone or fentanyl patch

Primary study parameters/outcome of the study:

Is methadone more effective than fentanyl in the treatment of pain in patients with head-and-neck cancer with respect to

1. significant pain relief (reduction of Numeric Rating Scale (NRS) of 50%) and
2. pain interference

Secondary study parameters/outcome of the study:

Is methadone superior to fentanyl in the treatment of pain in patients with head-and-neck cancer with respect to

1. time to achieve significant pain relief
2. side-effect profile?

DETAILED DESCRIPTION:
Study design The duration of the study will be 9 weeks. Patients will visit the outpatient clinic 5 times. Patients of MAASTRO clinic will be seen directly before or after the radiation therapy. No extra visits will be necessary.

T= -1: - informed consent

* sort of pain (DN4)
* randomisation

T = 0 - questionnaire 1: demographic variables, disease specific variables, BPI, side effect questions, HADS, QoL

* explain and provide the pain sheet
* start methadone 2 x 2,5 mg or fentanyl patch 12 μg/uur
* breakthrough medication: 50 µg fentanyl nose spray or fentanyl stick 400 µg till 6x/day

T=1 - questionnaire 2: BPI, side effect questions, global perceived effect

1 week - review pain sheet on pain and total rescue doses

* if necessary increase dose strong opioid with 50%

T=2 - questionnaire 2: BPI, side effect questions, global perceived effect 3 weeks - review pain sheet on pain and total rescue doses

* if necessary increase dose strong opioid with 50%
* if necessary decrease dose strong opioid with 30%

T=3 - questionnaire 2: BPI, side effect questions, global perceived effect 5 weeks - review pain sheet on pain and total rescue doses

* if necessary increase dose strong opioid with 50%
* if necessary decrease dose strong opioid with 30%

T = 4 - questionnaire 3: BPI, side effect questions, global perceived effect, QoL

* if necessary increase dose strong opioid with 50%
* if necessary decrease dose strong opioid with 30%

ELIGIBILITY:
Inclusion Criteria:

* opioid naive patients with histological proven head-and-neck cancer and (partly) neuropathic pain with a NRS score of =/> 4

Exclusion Criteria:

* age under 18
* not being able to read or fill in the questionnaires
* recent operation (less than 7 days)
* women of childbearing potential not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
significant pain relief (reduction of Numeric Rating Scale (NRS) of 50%) | 9 weeks

SECONDARY OUTCOMES:
time to achieve significant pain relief | 9 weeks
side-effect profile | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, MD, PhD, Study Chair — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands